CLINICAL TRIAL: NCT05320237
Title: Upper Limb Rehabilitation Using Immersive Virtual Reality for People With Multiple Sclerosis; a Feasibility Trial
Brief Title: Immersive Virtual Reality for Upper Limb Rehabilitation in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Collaborators: MS Society, UK (Unknown); NHS Lanarkshire (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22/VRMS/115
Record Dates: First submitted 2022-03-10; First posted 2022-04-11 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Rehabilitation; Virtual reality
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Intervention (Experimental): Eight weeks of two 30 minute sessions using virtual reality with the upper limb exercise games.
  Interventions: Other: Immersive Virtual Reality Intervention
- Control Group (No Intervention): Participants will be asked to continue with their usual care independent of this study.

INTERVENTIONS:
Other: Immersive Virtual Reality Intervention — Eight week intervention with two sessions a week. Each session will be 30 minutes in duration and will involve participants partaking in VR and such games include targeting individual finger movement (playing piano); grasp and release and one game (catching falling stars) includes holding a controller for elbow flexion and extension (Whack-a-mole).
  Arms: Virtual Reality Intervention

SUMMARY:
Virtual reality (VR) has reported benefits of engagement, immersion, and motivation in rehabilitation and has been proposed to be a solution for long-term engaging rehabilitation methods. However, the use of VR within the multiple sclerosis (MS) population is not widely investigated, and even less with regards to upper limb function. The main aim of this study is to assess the feasibility of using the Oculus Quest VR headset and games for improving upper limb function within the MS population. Recruited people with MS will be randomly assigned to either an eight week intervention using VR games that have been designed by co-production with people with MS and MS-specialists; or to a control group of usual care. All participants will undertake testing at baseline, four weeks and eight weeks for multiple outcomes measures related to upper limb and motor function. After completion of the intervention, participants who undertook VR intervention will complete a survey regarding the usability of the games, and some individuals will be invited to interviews to express their experience of using VR and any suggestions for improvement for potential future trials.

DETAILED DESCRIPTION:
The aim of this study is to investigate the feasibility of an eight-week intervention of co-produced virtual reality (VR) games delivered using the Oculus Quest for improving the upper limb function of people with MS. This study is also a randomised controlled trial with two arms, one group will undergo the intervention using VR and the other will be a control group.

This study aims to recruit up to 30 people with MS who have some degree of self-reported upper limb mobility difficulties from MS clinics in NHS Lanarkshire and MS Revive, a third sector in Glasgow. Participants will be randomly allocated to a group: an eight week intervention study using VR and exercise games or a control group of usual care. All groups will have assessments at baseline, week 4 and week 8. However, only the VR intervention group will undertake the USE questionnaire and only a select number of participants in the VR group will participate in the semi-structured interviews.

The VR intervention group will involve participants travelling to a research site twice a week for eight weeks and each session will be approximately 30 minutes. This 30-minute intervention will include participating in game play and the participant using the game's interface (e.g. navigating through menus, selecting which games to play). The games for the intervention will involve facilitating and replicating upper limb movements: pushing buttons for the interface; individual finger movement; grasp and release and one game includes holding a controller for elbow flexion and extension (see table). The intervention group will undergo exercises in a fully immersive VR environment using the Oculus Quest VR headsets. For health and safety reasons participants will complete their programme whilst seated.

The control group will not receive a specific exercise programme but will be asked to continue with their usual care, which could generally include any ongoing physiotherapy or occupational therapy support or none whatsoever. Any ongoing physiotherapy or occupational therapy (NHS or non-NHS) will be recorded, detailing the exercises and frequency. After completion of the week 8 assessment, participants within the control group will be offered the opportunity to take part in a 30-minute session trialling the VR games.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of multiple sclerosis.
* Degree of self-reported hand or upper limb impairment which interferes with some activities of daily living (ADL) (e.g. dressing, eating, grooming).
* Objective upper limb impairment, in at least one hand, as determined by a Nine Hole Peg Test (see Section Outcome Measures) of 2 standard deviations of more above the published normative values depending on age and sex.
* Must be able to travel to a research site.

Exclusion Criteria:

* If they have had a relapse in the last three months
* Subjective cognitive problems resulting in them being unable to use the equipment or participate in virtual reality.
* Visual problems such that they cannot see the visual display within the headset (this does not include participants who have glasses that are enough to correct eyesight issues)
* Have a current eye infection.
* Have any significant co-existing neurological or orthopaedic conditions affecting the upper limb.
* Are unable to understand verbal or written explanations of the study or are unable to speak or understand English.
* Individuals who are currently enrolled in any clinical trials will be excluded, but those who have previously taken part in research and other trials will be eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-06-26 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Recruitment Rates | First 5 months of study.
  Recording the number of participants: identified and approached; number of participants that meet eligibility criteria or are excluded and record reasons for exclusion; number of participants that agree to take part in the study.
Number of intervention sessions completed by participants | Through the intervention period of 6 months.
  Measured by recording the amount of VR sessions completed and the duration of these for each participant.
Recording the number of drop out rates from participants | Through the intervention period of 6 months.
  Measured by recording the amount of participants from both groups dropping out of the study.
Acceptance of being assigned to the control arm | Week 8 of intervention.
  Asking participants in the control arm if they accept being in this group rather than the intervention group.
Reporting adverse effects from intervention. | Through the intervention period of 6 months.
  Recording the number and type of adverse effects experienced by the participants from the intervention, either during or immediately following the VR intervention.
Rate of completion of secondary outcomes | Through the intervention period of 6 months.
  Recording if participants are able to complete the upper limb related outcomes.

SECONDARY OUTCOMES:
Nine Hole Peg Test | Baseline, Week 4, Week 8
  Measurement of hand dexterity.
ABLIHAND questionnaire | Baseline, Week 4, Week 8
  Self-reported questionnaire regarding their ability to perform activities of daily living that requires upper limb function. It has a maximum score of 46 and the lower the score, the poorer the functional ability.
Hand grip strength via Jamar dynamometer | Baseline, Week 4, Week 8
  Measurement of hand grip strength.
Action Research Arm Test (ARAT) | Baseline, Week 4, Week 8
  Measurement of ability of handling objects and other general upper limb movements.
The spasticity-related quality of life tool (SQoL-6D) | Baseline, Week 4, Week 8
  Self-reported questionnaire regarding how spasticity of their upper limb affects their quality of life. There are 7 domains and the participant has to tick which statement they believe is most appropriate to their spasticity within the last 7 days.
USE questionnaire | Week 8
  Questionnaire regarding the user's opinion on the usefulness, satisfaction and ease of use of the developed software. There are 30 questions using a 7-point Likert scale the participant must rate how strongly they agree or disagree with the statements regarding the software.
Semi-structured interviews | Week 9
  Interviews to explore the participant's experience with the virtual reality intervention, any issues encountered and suggested improvements for future studies using the games or virtual reality.

CONTACTS AND LOCATIONS:
Locations (1):
- Amy Webster, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to share participant data to anyone outside the research team, however the results of this study will be reported and planned publication after the study is completed with anonymised data.